CLINICAL TRIAL: NCT02707510
Title: A Randomized Controlled Trial to Strengthen Existential Resiliency Among Women With Metastatic Cancer
Brief Title: A Trial to Strengthen Existential Resiliency Among Women With Metastatic Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Arash Asher, MD, Director, Cancer Survivorship & Rehabilitation, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00043233
Record Dates: First submitted 2016-03-09; First posted 2016-03-14 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Breast Neoplasms; Neoplasm Metastasis
Keywords: logotherapy; cognitive behavior therapy; metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Arm (Experimental): Patients in the intervention group will be provided with all programmatic materials (including copies of power point presentations, copies of reading texts, and audio CDs) and classes will be held in group format, with a maximum of 9 participants per group. Classes will meet weekly, in a group, and at a set time. All classes will be facilitated jointly by the two Co-PIs. All participants will complete surveys before class, during class, at the end of class, 1 month after the end of class, 6 months after the end of class and 1 year after the end of the class. Additionally, those randomized to the intervention group will be asked to attend a 1 time focus group 1 week after the end of the class.
  Interventions: Other: Growing Resiliency And CouragE with Cancer™ (GRACE)
- Control Arm (No Intervention): Patients in the control group will be asked to complete surveys at: baseline, 6 weeks after baseline (T1), and 1 month after T1. After T1, the control group will off study and will be permitted to attend the next available GRACE course.

INTERVENTIONS:
Other: Growing Resiliency And CouragE with Cancer™ (GRACE) — GRACE is a 6 week curriculum which includes themes illustrated via PowerPoint slides with semi-structured delivery, video presentations, a variety of mindfulness meditation practices, and selected readings that serve to reflect and capture the theme for the week of the curriculum.
  Arms: Intervention Arm

SUMMARY:
The investigators group has piloted a 6-week psycho-educational program, Growing Resiliency And CouragE with Cancer™ (GRACE), that bring together a variety of strategies and experiences from an inter-professional perspective to mitigate distress among patients with an advanced cancer diagnosis. GRACE is a six-session, empirically anchored intervention emphasizing a Logotherapy (Existential Therapy) and Cognitive-Behavioral Therapy approach involving psycho-education and process-oriented experiences. The curriculum includes themes illustrated via PowerPoint slides with semi-structured delivery, video presentations, a variety of mindfulness meditation practices, and selected readings that serve to reflect and capture the theme for the week of the curriculum.

ELIGIBILITY:
Inclusion Criteria:

* Women with metastatic cancer with a minimum prognosis of 3 months
* Existential or spiritual concerns
* Reasonable medical stability as assessed by the evaluating physician
* Commits to attending 5/6 of the GRACE classes
* English speaking
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Unstable psychiatric disorder that would detract from a group program (i.e. severe depression/anxiety not controlled medically, volatile personality disorders)
* Cognitive impairment or cognitive linguistic impairment (i.e., aphasia) that would interfere with a group program.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
GRACE's Impact on Existential Distress (measured by survey) | Baseline to 6 weeks after baseline

SECONDARY OUTCOMES:
GRACE's Impact on Existential Distress (measured by survey) | Baseline to 10 weeks after baseline
GRACE's Impact on anxiety (measured by survey) | Baseline to 6 weeks after baseline
GRACE's Impact on anxiety (measured by survey) | Baseline to 10 weeks after baseline
GRACE's Impact on depression (measured by survey) | Baseline to 6 weeks after baseline
GRACE's Impact on depression (measured by survey) | Baseline to 10 weeks after baseline
GRACE's Impact on hopelessness (measured by survey) | Baseline to 6 weeks after baseline
GRACE's Impact on hopelessness (measured by survey) | Baseline to 10 weeks after baseline
GRACE's Impact on loneliness (measured by survey) | Baseline to 6 weeks after baseline
GRACE's Impact on loneliness (measured by survey) | Baseline to 10 weeks after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Arash Asher, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Asher A, Shirazipour CH, Capaldi JM, Kim S, Diniz M, Jones B, Wertheimer J. A 6-Week Program to Strengthen Resiliency Among Women With Metastatic Cancer: A Randomized Clinical Trial. Oncologist. 2023 Aug 3;28(8):e669-e682. doi: 10.1093/oncolo/oyad091. PMID 37104871